CLINICAL TRIAL: NCT04518605
Title: Breakfast for Young Females - the Importance of Breakfast Type
Brief Title: Breakfast for Young Females
Acronym: NyStart2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other); Sygekassernes Helsefond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: NyStart2
Record Dates: First submitted 2020-08-10; First posted 2020-08-19 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2021-07

CONDITIONS: Overweight and Obesity; Overweight Adolescents; Metabolic Disease
Keywords: Dairy protein; Breakfast content; body composition; Muscle strength; Gut microbiota/microflora; Dietary recommendations; Exercise training
MeSH Terms: conditions — Overweight; Obesity; Metabolic Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low protein breakfast (Experimental): Subject will eat a low protein breakfast and maintain their habitual physical activity.
  Interventions: Dietary Supplement: Low protein breakfast
- High protein breakfast (Experimental): Subject will eat a high protein breakfast and maintain their habitual physical activity.
  Interventions: Dietary Supplement: High protein breakfast
- Low protein breakfast and exercise training (Experimental): Subject will consume a low protein breakfast (bread, jam, juice) and and participate in organized exercise-training three times per week (and maintain habitual physical activity)
  Interventions: Dietary Supplement: Low protein breakfast; Other: Exercise training
- High protein breakfast and exercise training (Experimental): Subject will consume a high protein dairy breakfast (300 g high protein yoghurt (skyr) with oats) and and participate in organized exercise-training three times per week (and maintain habitual physical activity)
  Interventions: Dietary Supplement: High protein breakfast; Other: Exercise training

INTERVENTIONS:
Dietary Supplement: Low protein breakfast — Low protein yoghurt containing approx. 2 g protein per 100 g. Participants will be asked to consume ~60 g bread, 20 g jam and 250 ml juice for breakfast.
  Arms: Low protein breakfast; Low protein breakfast and exercise training
Dietary Supplement: High protein breakfast — High protein yoghurt containing approx. 10 g protein per 100 g. Participants will be asked to consume 300 g (=3 dl) yoghurt with 40 g oats for breakfast.
  Arms: High protein breakfast; High protein breakfast and exercise training
Other: Exercise training — Participants will be asked to participate in organized exercise training 3 times per week.
  Arms: High protein breakfast and exercise training; Low protein breakfast and exercise training

SUMMARY:
Investigators will test the health effects of eating a dairy-based protein-rich breakfast or isocaloric breakfast and performing regular physical exercise training for 12 weeks in young overweight women (2 x 2 factorial design). Measurements of body composition, physical fitness, metabolic health parameters, faeces and urine metabolites, and food diary will be collected.

DETAILED DESCRIPTION:
The study is a 2×2-factorial randomized controlled trial with 4 study arms. One-hundred (100) subjects will be randomly allocated to eat breakfast consisting of high-protein yoghurt (300g/day) with oats or an isocaloric breakfast consisting of bread, jam and juice matched for fat and fiber content and to either exercise 3x per week or maintain habitual physical activity for 12 weeks. Measurements and biological sampling will be performed at baseline, half way (some parameters only) and at the end of the intervention period.

The primary outcome will be fat mass and fat free mass determined by DXA. The investigators will also measure effects on weight, waist, health-related blood parameters, muscle function, physical activity, habitual food intake and metabolites in faeces, urine and blood.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 25
* Regular exercise < 1 hour per week

Exclusion Criteria:

* illness and use of medication affecting the study outcomes
* allergy towards milk and yoghurt
* weightloss/gain >5kg the last 6 months
* dieting
* eating disorder
* pregnancy
* breast feeding
* unable to speak and understand danish

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Fat mass in grams | 12 weeks
  Measured by dual energy x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Change in Fat free mass in grams | 12 weeks
  Measured by dual energy x-ray absorptiometry (DXA)
Change in Lean body mass in grams | 12 weeks
  Measured by dual energy x-ray absorptiometry (DXA)
Change in Height (cm) | 12 weeks
  by stadiometer
Change in weight (kg) | 12 weeks
  Tanita Scale
Change in BMI (m^2/kg) | 12 weeks
  Measured by height in meters and weight in kg
Change in Waist circumference (cm) | 12 weeks
  by tape
Change in HbA1c | 12 weeks
  by fasting blood sample
Change in high density lipoprotein cholesterol (HDL cholesterol) | 12 weeks
  by fasting blood sample
Change in low density lipoprotein cholesterol (LDL cholesterol) | 12 weeks
  by fasting blood sample
Change in triacylglycerol (TG) | 12 weeks
  by fasting blood sample
Change in total cholesterol | 12 weeks
  by fasting blood sample
Change in glucose | 12 weeks
  by fasting blood sample
Change in insulin | 12 weeks
  by fasting blood sample
Change in glucose tolerance (area under the curve) | 12 weeks
  measured by a two hour oral glucose tolerance test
Change in glucose peak | 12 weeks
  measured by a two hour oral glucose tolerance test
Change in fitness (estimated VO2-max) | 12 weeks
  Measured by Åstrand two-step bike test
Change in maximal hand grip strength | 12 weeks
  Measured by hand held dynamometer
Change in maximal arm strength | 12 weeks
  Measured by costummade dynamometer
Change in maximal jump height | 12 weeks
  Measured by squat jump with linear encoder
Change in systolic and diastolic blood pressure | 12 weeks
  by standard blood pressure apparatus

OTHER OUTCOMES:
Change in physical activity | 12 weeks
  by accelerometry
Changes in dietary intake | 12 weeks
  by 4-day dietary registration
Changes in calcium and supplement intake | 12 weeks
  by a standard, validated food frequency questionnaire.
Change in gut microflora | 12 weeks
  by bacterial determination of faeces
Changes in faeces pH | 12 weeks
  by pH determination of faeces
Changes in urine metabolites | 12 weeks
  To evaluate the effect of the intervention on metabolism through a metabolomic approach. Urine samples will be collected to perform a metabolomics analysis by mass spectroscopy.
Changes in faeces metabolites | 12 weeks
  To evaluate the effect of the intervention on the metabolism through a metabolomic approach. Faeces samples will be collected to perform a metabolomics analysis by mass spectroscopy.
Changes in blood metabolites | 12 weeks
  To evaluate the effect of the intervention on metabolism through a metabolomic approach. Blood samples will be collected to perform a metabolomics analysis by mass spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, Assoc Prof, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dalgaard LB, Thams L, Skovgaard Jensen J, Jorgensen AA, Breenfeldt Andersen A, Gejl KD, Bertram HC, Hansen M. No effects of high- v. low-protein breakfast on body composition and cardiometabolic health in young women with overweight: the NewStart randomised trial. Br J Nutr. 2025 Jan 14;133(1):126-135. doi: 10.1017/S0007114524003015. Epub 2024 Nov 26. PMID 39587799